CLINICAL TRIAL: NCT02995746
Title: Intravitreal Dexamethasone Implant for Persistent Macular Thickening and Edema After Vitrectomy for Epiretinal Membrane: A Pilot Study
Brief Title: Intravitreal Dexamethasone Implant for Persistent Macular Thickening and Edema After Vitrectomy for Epiretinal Membrane
Acronym: DEMO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to lack of drug efficacy. 2017 study did not show benefit.
Sponsor: Wills Eye (Other)
Collaborators: Mid Atlantic Retina (Other)
Responsible Party: Principal Investigator, Allen C. Ho, MD, MD, Wills Eye
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-475
Record Dates: First submitted 2016-09-14; First posted 2016-12-16 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Macular Edema; Epiretinal Membrane; Vitrectomy
MeSH Terms: conditions — Macular Edema; Epiretinal Membrane | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0.7mg dexamethasone intravitreal implant (Experimental): Single intravitreal implantation of 0.7mg dexamethasone with a six month follow up period
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — * On study visit #1 all patients will have a SD-OCT scan and measurement of baseline visual acuity. All patients will receive the 0.7mg dexamethasone intravitreal implant
  * Subsequent follow-up visits will be at 1 month, 2 months, 3 months, 4 months, 5 months, and 6 months after intravitreal injection of dexamethasone implant
  * Each visit will consist of measurement of visual acuity, intraocular pressure, dilated fundoscopic examination, and SD-OCT scan
  * Anticipated duration of the study: 6 months
  Other Names: Ozurdex

SUMMARY:
This study seeks to evaluate the effect of the intravitreal 0.7mg dexamethasone implant on central macular thickness and visual acuity in those patients with persistent macular edema after pars plana vitrectomy for epiretinal membrane.

DETAILED DESCRIPTION:
Macular edema is a relatively common occurrence after pars plana vitrectomy. Kim et al described that 47% of eyes undergoing vitrectomy for epiretinal membrane, macular hole, or vitreous hemorrhage had evidence of macular thickening on optical coherence tomography scan.1 Post-vitrectomy macular edema can limit potential visual acuity gain from removal of a symptomatic epiretinal membrane. Typical treatment of post-operative macular edema consists of topical non-steroidal anti-inflammatory drugs (NSAIDs) and topical corticosteroids; however, there are still resistant cases with refractory macular thickening.

The dexamethasone intravitreal implant (Ozurdex; Allergan, Irvine, CA) is currently FDA-approved for the treatment of posterior uveitis as well as macular edema secondary to retinal vein occlusion and diabetic retinopathy. Furino et al reported a retrospective series describing how a single injection of the 0.7mg dexamethasone intravitreal implant resulted in a substantial increase in best-corrected visual acuity (BCVA) and a decrease in central macular thickness (CMT) on spectral-domain optical coherence tomography (SD-OCT) in 8 patients with persistent macular thickening after pars plana vitrectomy for epiretinal membrane. There has been no prospective study evaluating the efficacy of this pharmacologic agent in this setting.

As such, the purpose of this study is to prospectively evaluate the effect of the intravitreal 0.7mg dexamethasone implant on CMT and BCVA in those patients with persistent macular edema after pars plana vitrectomy for epiretinal membrane.

The results of this study will help delineate whether the intravitreal dexamethasone implant has efficacy in improving CMT and/or visual acuity in those patients with refractory macular thickening after pars plana vitrectomy for epiretinal membrane.

ELIGIBILITY:
Inclusion Criteria:

1. Patient of the Wills Eye Institute Retina service, including all Mid-Atlantic Retina offices
2. Volunteer patients age 18 years and older
3. Healthy enough to participate in the study
4. Willing and able to consent to participation in the study
5. History of pars plan vitrectomy for symptomatic epiretinal membrane at least 3 months prior to study enrollment date
6. BCVA of 20/40 or worse
7. CMT of at least 400 micrometers with or without cystoid macular edema on SD-OCT
8. Prior treatment with topical NSAIDs without resolution of macular thickening or visual acuity improvement

Exclusion Criteria:

1. Advanced glaucoma (cup-disc ratio of 0.8 or greater)
2. History of glaucoma filtering or tube shunt implant surgery
3. Steroid responsive intraocular hypertension
4. Diabetic retinopathy
5. History of uveitis
6. Use of systemic or intraocular corticosteroids
7. Active or suspected ocular or periocular infections
8. Other confounding intraocular pathology

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
Mean central macular thickness (CMT) on SD-OCT at 1 month, 3 months, and 6 months after intravitreal injection of dexamethasone implant | Change in mean macular thickness baseline at 6 months

SECONDARY OUTCOMES:
Visual acuity | Change in visual acuity baseline at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Allen C Ho, MD, Principal Investigator — Mid Atlantic Retina
Locations (1):
- Mid Atlantic Retina, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No